CLINICAL TRIAL: NCT06570694
Title: A Mobile Ecological Momentary Intervention for Reducing Experiential Avoidance in the Context of Rumination: Protocol for a Randomised-Controlled Trial
Brief Title: RCT Protocol for 'OverThinking': A Mobile EMI for Reducing Experiential Avoidance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Collaborators: Polish Japanese Academy of Information Technology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SWPS-ECL-WKEB90/11/2023
Record Dates: First submitted 2024-08-19; First posted 2024-08-26 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Depression; Anxiety; Rumination
Keywords: Rumination; Experiential Avoidance; Depression; Anxiety; Ecological momentary intervention
MeSH Terms: conditions — Depression; Anxiety Disorders; Rumination Syndrome

STUDY DESIGN:
Intervention Model Description: Four arm parallel-group trial:
  (1) intervention condition (therapist support); (2) intervention condition (no therapist support); (3) Partial intervention (daily sampling and emotion valuation questions); (4) Control group (only daily sampling questions).
Who Masked: Participant
Masking Description: Participants will be allocated to condition via a random number generator and will be provided with trial instructions pertaining only to their allocated condition. Trial participants will not be provided with any information relating to the remaining three conditions in the trial until the 1-month follow-up period has elapsed.
  The member of the research team responsible for analysing the data will additionally be blinded to the allocation of participants. This will be anonymised for them in the dataset without accompanying explanatory label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Intervention Group 1: Concurrent Therapist Support (Experimental): Participants will receive the four-week intervention via the mobile application. This will be supplemented with asynchronous written support from a CBT practitioner (qualified or after the second year of their training) via WhatsApp and will be available twice a week to relevant participants at specific times predetermined by the therapist. Participants will be available to utilise this support but will not be directed to do so. Participants in this condition will, as part of their use of the application, participate in providing daily sampling, which includes emotion valuation questions.
  Interventions: Behavioral: OverThinking
- Intervention Group 2: No Concurrent Therapist Support (Experimental): Participants will receive the four-week intervention via the mobile application. No concurrent therapist support will be provided in this group. Participants in this condition will, as part of their use of the application, participate in providing daily sampling, which includes emotion valuation questions.
  Interventions: Behavioral: OverThinking
- Partial Intervention (No Intervention): Partial intervention group: This group will not receive the four-week mobile intervention, but will participate in providing daily sampling (via web-based form), which includes emotion valuation questions.
- Control (No Intervention): Control group: This group will not receive the four-week mobile intervention, but will participate in providing daily sampling (via web-based form) - this does not include emotion valuation questions.

INTERVENTIONS:
Behavioral: OverThinking — OverThinking is a mobile application ecological momentary intervention for iOS and Android, which has been designed for the reduction of experiential avoidance in rumination. The application primarily consists of psychoeducation content and related exercises intended to be delivered over a four-week period. In order to examine the effectiveness of the application during the course of the intervention and to examine user-experiences of using the application for the purpose of rumination intervention, a number of self-report tools are embedded.
  Arms: Intervention Group 1: Concurrent Therapist Support; Intervention Group 2: No Concurrent Therapist Support

SUMMARY:
The goal of this trial is to examine whether a mobile app intervention for rumination can modify a maladaptive feature of repetitive negative thinking (RNT) - this is understood by the link between daily RNT and well-being, depressive and anxiety symptoms.

The main questions it aims to answer are:

1. If the intervention can modify the maladaptive feature of repetitive negative thinking - the investigators anticipate the link between daily rumination and maladaptive outcomes (poorer wellbeing, higher depressive/anxious symptoms) will be weaker in the intervention groups.
2. By examining (1) above, to confirm the role played by avoidance in repetitive negative thinking.
3. By splitting the intervention condition into two groups (one receiving concurrent support from a therapist, one not), to evaluate if interventions such as these might be enhanced by therapist support.
4. To examine if the impact of the intervention on depressive and anxious symptoms might be mediated by changes in beliefs regarding emotions (e.g. the valuation of negative emotions).

Researchers will compare across four groups to examine the above effects:

(1) intervention condition (therapist support); (2) intervention condition (no therapist support); (3) Partial intervention (daily sampling and emotion valuation questions); (4) Control group (only daily sampling questions).

Participants will:

* Be requested to participate in a four-week intervention, providing daily assessments of depressive and anxiety symptoms, affect, repetitive negative thinking, and rumination outcomes.
* Use a mobile application during the intervention period, which has been designed by the research team (intervention groups), or provide daily assessment scores only (control groups).
* Be assessed at pre-intervention (all groups), post-intervention (all groups), 1-month follow-up (all groups), and 3-month follow-up (intervention groups only).

DETAILED DESCRIPTION:
The trial aims to examine whether a mobile application-based intervention for experiential avoidance in the context of rumination can modify a maladaptive feature of repetitive negative thinking (RNT) - this is understood by the link between daily RNT and well-being, depressive and anxiety symptoms.

The main questions which the trial aims to answer are as follows:

1. If the intervention can modify the maladaptive feature of repetitive negative thinking - the investigators anticipate the link between daily rumination and maladaptive outcomes (poorer wellbeing, higher depressive/anxious symptoms) will be weaker in the intervention groups.
2. By examining (1) above, to confirm the role played by avoidance in repetitive negative thinking.
3. By splitting the intervention condition into two groups (one receiving concurrent support from a therapist, one not), to evaluate if interventions such as these might be enhanced by therapist support.
4. To examine if the impact of the intervention on depressive and anxious symptoms might be mediated by changes in beliefs regarding emotions (e.g. the valuation of negative emotions).

Researchers will compare across four groups to examine the above effects:

(1) intervention condition (therapist support); (2) intervention condition (no therapist support); (3) Partial intervention (daily sampling and emotion valuation questions); (4) Control group (only daily sampling questions).

The trial comprises of a four-arm, parallel group randomised-controlled trial (RCT). Participation lasts approximately 2 months (including eligibility screening and random allocation to condition (random number generator), a four-week intervention period delivered via the mobile application and supplemented with daily assessments, post-intervention assessments, and 1-month follow-up (wherein the app will remain available for self-directed use without daily sampling), concluding with follow-up assessments and measurement of any engagement with the application during this period.

At the point of 1-month follow-up, participants previously allocated to the control groups will receive access to the application (without the feature of daily sampling) and will be provided with guidance on using the intervention content. While a 3-month follow-up assessment of intervention participants is planned, the 1-month interval allows for control participants to access intervention content without being subject to extensive waitlist delay. Active control groups have been chosen to not artificially inflate comparisons with outcomes in the intervention conditions.

Analysis:

Analysis of changes in outcomes across pre-, post- and follow-up-measures (PTQ, EBQ, PBRS, NBRS, HADS, CAQ, and BEAQ) across all four conditions will be conducted using mixed-design ANOVA.

Additionally for all conditions, multilevel models (daily observations on level 1 nested in participants on level 2) will be used on daily sampling data to assess the links between avoidance and mood and between rumination and mood, and to determine if each of these links is moderated by condition. Participants respond to these items once daily in the evening, in response an in-app reminder alert (the time of the alert can be determined by the participant). All daily sampling items have been provided in the 'Measures' section.

Mixed-design ANCOVA will be used for the two intervention groups to examine if time spent engaging with the application content acts as a covariate in intervention outcomes (PTQ, EBQ, PBRS, NBRS, HADS, CAQ, and BEAQ).

Finally, ongoing development of the application will be assisted using in-app user-feedback data obtained via CORTO implementation (three items with gather a combination of quantitative and qualitative data [Lukka et al,. 2024]). This data will be coded deductively using the process outlined by Saldana (2016) and using the four categories identified by Lukka et al. (2024) as high-level guidance ((1) contextual use, (2) interaction-elicited emotional experience, (3) usability, and (4) technical issues.), with more detailed coding examined as subdomains.

ELIGIBILITY:
Inclusion Criteria:

- Self-reporting problems with repetitive negative thinking.

Exclusion Criteria:

* Aged below 18 years at the commencement of the trial.
* Currently in receipt of any form of psychotherapy.
* Currently in receipt of any form of psychiatric medication.

Note: Participants who hold a psychiatric diagnosis will not be excluded from the trial provided they meet the inclusion criterion and do not meet any of the exclusion criteria listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Perseverative thinking as measured by the Perseverative Thinking Questionnaire (PTQ) | Two months (4-week intervention plus 1-month follow-up)
  The PTQ is a 15-item self-report measure, which assesses the main characteristics of repetitive negative thinking (1: core features - 9 items, 2: unproductiveness - 3 items, 3: capturing mental capacity - 3 items. Responses are recorded on a scale of '0' ('never') to '4' ('almost always').
Beliefs about emotions as measured by the Emotion Beliefs Questionnaire EBQ | Two months (4-week intervention plus 1-month follow-up)
  The EBQ is a 16-item self-report questionnaire intended to measure the controllability of emotions and respondent beliefs about the usefulness of emotions. Respondents answer using a 7-point Likert scale ranging from 1 (totally disagree) to 7 (totally agree), with high scores indicating a belief that emotions are uncontrollable and/or useless.
Metacognitive beliefs about rumination using PBRS/NBRS | Two months (4-week intervention plus 1-month follow-up)
  This is comprised of two sub-scales (positive beliefs: 9-items, negative beliefs: 13-items) measuring metacognitive beliefs of depressive rumination. Respondents rate the extent to which they agree with each of the items using a 4-point Likert-type scale ranging from 1 (do not agree) to 4 (agree very much), with higher scores on each subscale indicating greater positive/negative belief accordingly.
Hospital Anxiety and Depression Scale (HADS) | Two months (4-week intervention plus 1-month follow-up)
  A measure of possible and probable presence of anxiety disorders and depression, comprising seven items for depression and seven items for anxiety. Respondents rate on a scale of 0-3 for each item, with higher total scores for each subdomain (anxiety, depression) indicating greater presence of the disorder. Thresholds are provided for determining the clinical presence of disorder as follows: 0-7 = Normal, 8-10 = Borderline abnormal (borderline case),11-21 = Abnormal (case)
Cognitive avoidance using the CAQ | Two months (4-week intervention plus 1-month follow-up)
  A 25-item measure of five worry-related cognitive avoidance strategies (thought suppression, thought substitution, distraction, avoidance of threatening stimuli, transformation of images into thoughts). The scale comprises five subscales, each containing five items, which represent individual cognitive avoidance strategies (avoidance of threatening stimuli, distraction, thought substitution, thought suppression, transformation of images into thoughts). Respondents answer on a five-point scale (1: not at all applicable, to 5: very applicable), with higher scores indicating greater presence of cognitive avoidance.
Experiential avoidance using the BEAQ. | Two months (4-week intervention plus 1-month follow-up)
  A 15-item short-version of the Multidimensional Experiential Avoidance Questionnaire, measuring EA content across six dimensions. Respondents provide answers to pre-determined statements along a 6-point Likert scale ('1': strongly disagree; to '6': strongly agree), with higher scores indicating a greater presence of experiential avoidance.
Daily Sampling Items (1: Repetitive Negative Thinking Items) | Once daily for 30 days
  Nine items relating to different dimensions of repetitive negative thinking derived from the scale by Rosenkrantz et al. (2020) (feelings, problems, past, future, duration, distress, repetitiveness, intrusiveness, uncontrollability). These are answered on a scale from 1-7 (1: "not at all", 7: "very much"), with a higher overall score indicating a greater presence of issues with repetitive negative thinking.
Daily Sampling Items (2: Depression) | Once daily for 30 days
  Three items developed from the scale by Krejtz et al. (2016), which ask the participant about their day (1: "very negative", 7: "very positive"), the extent to which they felt positive about themselves that day (1: "not at all", 7: "very much") and how they are feeling about tomorrow (1: "very negative", 7: "very positive"). Higher total scores indicate greater severity of difficulties with depression on that day.
Daily Sampling Items (3: Affect) | Once daily for 30 days
  Four closed-ended items adapted from Pe et al. (2013) (rated on a scale of 1: "not at all", to 7: "very much"), which ask the participant about the extent to which they felt nervous/anxious, sad, angry, and disgusted during the day. Additionally, an open-ended item is presented asking participants to 'Choose the emotion that you felt the strongest - what useful function could it have played for you today?'
Daily Sampling Items (4: Goals) | Once daily for 30 days
  Adapted from Moberly & Watkins (2010), participants are asked to enter a goal of importance to them during the day. Two follow-up questions then ask: 1) How important was this goal? (1: "not at all", 7: "very much"), and 2) To what extent did you manage to achieve this goal? (1: "not at all", 7: "very much")
Daily Sampling Items (5: Rumination Outcomes) | Once daily for 30 days
  Three items assessing the productivity of the individual's engagement in rumination, emotional discomfort resulting from rumination, and rumination-induced motivation during the day: 1) How productive was your rumination today? (1: "not at all", 7: "very much"), 2) How difficult/painful/comfortable was this reflection for you? (1: "not at all", 7: "very much"), and 3) Did it motivate you to take specific action? (1: "definitely not, 7: "definitely yes")

SECONDARY OUTCOMES:
Time spent using the application | During the 4-week intervention period and 1-month follow-up period
  The application has been designed to record the amount of time a user is active (and in which in-app exercises). This data is stored remotely and securely via Firebase. This data is password protected and access is limited to the individuals on the research team.

OTHER OUTCOMES:
Ongoing Application Development Feedback (CORTO) | During the 4-week intervention period and 1-month follow-up period
  Three items (two quantitative and two qualitative) collected following each in-app exercise, with the aim of providing real-time user-experience data to enable the ongoing development of the app. Items include: 1) Do you like using the application? (1: "not at all", 7: "very much"), 2) How would you rate the difficulty level of using the application? (1: "definitely too easy", 7: "definitely too difficult"), and 3) Would you like to share any thoughts about the app? (open-ended question).
  Data obtained via CORTO implementation will be coded deductively using the process outlined by Saldana (2016) and using the four categories identified by Lukka et al. (2024) as high-level guidance ((1) contextual use, (2) interaction-elicited emotional experience, (3) usability, and (4) technical issues.), with more detailed coding examined as subdomains.

CONTACTS AND LOCATIONS:
Overall Officials: Monika Kornacka, PhD, Principal Investigator — SWPS University

IPD SHARING:
Plan to Share IPD: Yes
Following the conclusion of the trial and the peer-reviewed publication of findings, data will be made available in anonymised form via the Open Science Framework.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become publicly available once the trial has concluded and once the outcomes have been published in a peer-reviewed outlet. The investigators do not anticipate any expiration date for the availability of this data once publicly disseminated.

REFERENCES:
- [Derived] Barnes S, Szastok M, Para M, Morawiec F, Grzeszczuk M, Wojcik S, Karpowicz B, Zinevych P, Jaskulska A, Kopec W, Kornacka M. A Mobile Ecological Momentary Intervention for Reducing Experiential Avoidance in the Context of Rumination: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 May 27;14:e66067. doi: 10.2196/66067. PMID 40424024